CLINICAL TRIAL: NCT04986995
Title: Open-label, Single-arm, Pilot Study to Evaluate the Effect of Opicapone 50 mg on Parkinson's Disease Patients With End-of-dose Motor Fluctuations and Associated Sleep Disorders
Brief Title: OpicApone Sleep dISorder
Acronym: OASIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-405; 2020-001176-15 (EudraCT Number)
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opicapone (Experimental): 50 mg hard capsules
  Interventions: Drug: Opicapone

INTERVENTIONS:
Drug: Opicapone — Oral administration, once daily, at least 1 hour before or after the last daily dose of L-dopa/DDCI
  Other Names: BIA 9-1067

SUMMARY:
The aim of this study is to To investigate in an exploratory manner the efficacy of 50 mg opicapone when administered with the existing treatment of levodopa (L-dopa) plus a dopa decarboxylase inhibitor (DDCI), in Parkinson's disease (PD) patients with end-of-dose motor fluctuations and associated sleep disorders

DETAILED DESCRIPTION:
This is an open-label, single-arm, multi-centre, interventional clinical study in PD patients with end-of-dose motor fluctuations and associated sleep disorders. The study consists of a 1-week screening period, a 6-week treatment period and 2 weeks of follow-up period. Expected duration of treatment for the individual patient is up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form and to comply with all aspects of the study.
2. Male or female patients aged 30 years or older.
3. Diagnosed with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria (2006) or according to MDS Clinical Diagnostic Criteria (2015).
4. Signs of "wearing-off" phenomenon (end-of-dose motor fluctuations) with average total daily OFF time while awake of at least 1.5 hours, excluding the early morning pre-first dose OFF, despite optimal anti-PD therapy (based on investigator's assessment).
5. Disease severity Stages I-III (modified Hoehn & Yahr staging) at ON.
6. Experiencing PD associated sleep disorders for at least 4 weeks prior to V1.
7. Total PDSS-2 score ≥ 18.
8. Treated with 3 to 8 intakes per day of L-dopa/DDCI (which may include a slow-release formulation), on a stable regimen for at least 4 weeks before V1.
9. In case of any other anti-PD treatment, it should be on a stable regimen for at least 4 weeks before V1, and not likely to need any adjustment until V4.
10. No change in the chronic treatment regimen within the last 4 weeks before V1 of the following medication: sedatives, hypnotics, anti-depressants, anxiolytics or other medications prescribed for the treatment of sleep disorders
11. For females: Postmenopausal for at least 2 years before V1, surgically sterile for at least 6 months before V1, or practicing an effective method of contraception until V4. Female patients who request to continue with oral contraceptives must be willing to use non-hormonal methods of contraception in addition during the course of this study.

    For males: Male patients who are sexually active with a partner of childbearing potential must use, with their partner, a condom plus an approved method of highly effective contraception during the treatment period until V4.
12. Have filled-in self-rating diary in accordance with the diary instructions and with ≤ 3 errors per day when awake, in the 3 days preceding V2a/V2b.
13. With at least 1.5 OFF hours per day, excluding the early morning pre-first dose OFF period (i.e. the time between wake-up and response to the first L dopa/DDCI dosage), as recorded in at least 2 of the 3 days in the self-rating diary for the 3 days preceding V2a/V2b.
14. Total PDSS-2 score ≥ 18.
15. Adequate compliance to relevant (PD and sleep disorders) concomitant medication during the screening period (based on the investigator's judgment).

Exclusion Criteria:

1. Non-idiopathic PD (atypical parkinsonism, secondary [acquired or symptomatic] parkinsonism, Parkinson-plus syndrome).
2. Severe and/or unpredictable OFF periods, according to investigator judgement.
3. Major/prominent non-PD-related sleep disorders (e.g. sleep apnoea or narcolepsy).
4. Treatment with prohibited medication: entacapone, tolcapone, monoamine oxidase (MAO) inhibitors (except selegiline up to 10 mg/day in oral formulation or 1.25 mg/day in buccal absorption formulation, rasagiline up to 1 mg/day or safinamide up to 100 mg/day), or antiemetics with antidopaminergic action (except domperidone) within the last 4 weeks before V1 or likely to be needed at any time until V4.
5. Treatment with apomorphine within the last 4 weeks before V1 or likely to be needed at any time until V4.
6. Previous or current use of opicapone.
7. Previous or planned (until the end of this study) L-dopa/carbidopa intestinal gel infusion, deep brain stimulation or stereotactic surgery (e.g. pallidotomy, thalamotomy).
8. Use of any other investigational product (IP), currently or within the 3 months (or within 5 half-lives of the IP, whichever is longer) before V1.
9. Past (within the past year) or present history of suicidal ideation or suicide attempts.
10. Current or previous (within the past year) alcohol or substance abuse excluding caffeine or nicotine.
11. Phaeochromocytoma, paraganglioma, or other catecholamine secreting neoplasms.
12. Known hypersensitivity to the excipients of IP (including lactose intolerance, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption).
13. History of neuroleptic malignant syndrome or non-traumatic rhabdomyolysis.
14. History of severe hepatic impairment (Child-Pugh Class C).
15. Previous history of psychosis or psychiatric disorders, including severe major depression.
16. Any medical condition that might place the patient at increased risk or interfere with assessments.
17. For females: Pregnant or breastfeeding.
18. Employees of the investigator, study centre, sponsor, clinical research organisation and study consultants, when employees are directly involved in this study or other studies under the direction of this investigator or study centre, and their family members.
19. Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Total score of Parkinson's Disease Sleep Scale - version 2 (PDSS-2) | Up to 6 weeks
  Parkinson's Disease Sleep Scale version 2 (PDSS-2) is a patient-completed clinical rating scale that assesses the frequency of sleep disturbances over the past week. Each question is scored between 0 ("never") and 4 ("very often"), and a total score is calculated by summing a patient's responses to each of the 15 questions (minimum 0 to maximum 60)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital da Senhora da Oliveira - Guimarães, E.P.E, Serviço de Neurologia, Guimarães, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trenkwalder C, Kohnen R, Hogl B, Metta V, Sixel-Doring F, Frauscher B, Hulsmann J, Martinez-Martin P, Chaudhuri KR. Parkinson's disease sleep scale--validation of the revised version PDSS-2. Mov Disord. 2011 Mar;26(4):644-52. doi: 10.1002/mds.23476. Epub 2011 Feb 10. PMID 21312275
- See also: Parkinson's disease sleep scale--validation of the revised version PDSS-2 — https://pubmed.ncbi.nlm.nih.gov/21312275/